CLINICAL TRIAL: NCT02977039
Title: Effect of a Nutrient Dense Plant Rich Diet on Glycemic Control in People With Type 2 Diabetes and Obesity
Brief Title: Effect of a Plant Rich Diet on in People With Type 2 Diabetes and Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Martin Abrahamson, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000321
Record Dates: First submitted 2016-11-20; First posted 2016-11-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus in Obese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NDPR diet (Experimental): Subjects randomized to the nutrient dense plant rich (NDPR) diet will eat foods with high micronutrient density, and favorable glycemic index. The diet is low in saturated fat, high in fiber, and rich in phytochemicals. Total caloric intake will range from 1600-2000/day based on individual needs. Foods include vegetables (30-70% of calories), fruits (15-20% of calories), Beans/Legumes (20-30% of calories), raw nuts and seeds (10-20% of calories), fish or fat-free dairy (twice weekly or less), poultry, eggs and oils (once weekly or less) and limited beef, cheese/milk, processed food and beef.
  Interventions: Other: NDPR diet
- USDA diet (Experimental): Subjects randomized to the healthy U.S.-Style pattern diet will eat the types and proportions of foods Americans typically consume, but in nutrient-dense forms and appropriate amounts. It is designed to meet nutrient needs while not exceeding calorie requirements and while staying within limits for overconsumed dietary components. Total caloric intake will range from 1600-2000/day based on individual needs. Foods include fruits, vegetables (dark green, red/orange, beans, and peas, starchy vegetables), grains (whole grains and refined grains), protein foods (meat, poultry, eggs, seafood, nuts, seeds and soy products), dairy, and oils.
  Interventions: Other: USDA healthy eating diet

INTERVENTIONS:
Other: NDPR diet — nutrient rich plant based diert
  Arms: NDPR diet
Other: USDA healthy eating diet — DASH diet
  Arms: USDA diet

SUMMARY:
The purpose of this study is to evaluate the effect of a nutrient dense plant rich (NDPR) diet compared to a standard USDA diet on glycemic control, inflammation, and cardiovascular risk in individuals with type 2 diabetes and overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18-75
2. Type 2 diabetes mellitus diagnosed > 6 months prior to screening visit according to American Diabetes Association criteria
3. HBA1c >7.5% but < 10%
4. BMI >25 kg/m2 ; >23 kg/m2 for Asian subjects but < 45 kg/m2
5. Stable weight (variation < 5 kg within 6 months of screening visit)
6. Ability to give informed consent
7. Ability to follow verbal and written instructions in English

Exclusion Criteria:

1. Active cardiac issues: history of myocardial infarction within 3 months of screening visit, unstable angina pectoris, or Class III or Class IV congestive heart failure
2. Persistent uncontrolled hypertension (BP > 160/100 mmHg on or off antihypertensive medication)
3. Active marijuana or intravenous drug use
4. Recent weight loss (> 5 kg within 6 months of the screening visit)
5. Inflammatory or irritable bowel disease (Crohn's Disease, Ulcerative Colitis, or IBS)
6. Celiac disease
7. Malignancy treated with chemotherapy within the past 1 year
8. Depression or psychosis requiring hospitalization within 1 year, or use of major antipsychotic or tranquilizer drugs (i.e. benzodiazepines)
9. Renal insufficiency (creatinine clearance < 30 ml/min)
10. Transaminases > 2x above the normal range
11. Pregnancy within 6 months of the screening visit
12. Lactation
13. History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling
14. History of alcohol abuse within the past 5 years
15. Vegetarian/Vegan diet
16. Dairy Allergy/Intolerance
17. Anemia, including iron deficient and megaloblastic
18. Vitamin B12 deficiency
19. Leber's disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | change at 1, 3, 6, 9, 12 months
  A1C and finger stick blood sugar levels

SECONDARY OUTCOMES:
body weight | change at 1, 3, 6, 9, 12 months
body composition | change at 1,3,6,9, 12 months
  DXA scan
hepatic steatosis | baseline, 1, 3, 6, 9, 12 months
  MRspectroscopy
inflammatory markers | change at, 1, 3, 6, 9, 12 months
  serum inflammatory markers
quality of life | change at, 1, 3, 6, 9, 12 months
  validated questionnaired

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data with other researchers